CLINICAL TRIAL: NCT06069804
Title: Triamcinolone Acetonide as an Adjuvant to Pre-emptive Scalp Infiltration for Relief of Post-craniotomy Pain in Adults
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Beijing Tiantan Hospital (Other)
Responsible Party: Principal Investigator, Fang Luo, Director of Department of Pain Management, Beijing Tiantan Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: KY 2018-034-02-4
Record Dates: First submitted 2023-09-24; First posted 2023-10-06 (Actual); Last update posted 2024-04-03 (Actual); Status verified 2024-04

CONDITIONS: Pain, Postoperative
Keywords: Postoperative Pain;; Post-Craniotomy; Pre-emptive Scalp Infiltration; Ropivacaine; Triamcinolone Acetonide
MeSH Terms: conditions — Pain, Postoperative

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- The TR group (Experimental): The respective drugs to be used for incision-site infiltration were prepared by an independent study investigator in the two groups: Participates will receive peri-incisional scalp infiltration with10 mg triamcinolone acetonide, 150 mg ropivacaine diluted to a total volume of 30 mL in 0.9% saline . The concentration of ropivacaine was 0.5% in both groups. The anesthesia protocol and monitoring were standardized for all patients. Monitoring, including blood pressure (BP), heart rate (HR), 5-lead electrocardiography (ECG), peripheral oxygen saturation (SpO2) and bispectral index (BIS) were continuously performed.
  Interventions: Drug: The TR group
- The R group (Active Comparator): The respective drugs to be used for incision-site infiltration were prepared by an independent study investigator in the two groups: Participates will receive peri-incisional scalp infiltration with 150 mg ropivacaine diluted to a total volume of 30 mL in 0.9% saline in the control group. The concentration of ropivacaine was 0.5% in both groups. The anesthesia protocol and monitoring were standardized for all patients. Monitoring, including blood pressure (BP), heart rate (HR), 5-lead electrocardiography (ECG), peripheral oxygen saturation (SpO2) and bispectral index (BIS) were continuously performed.
  Interventions: Drug: The R group

INTERVENTIONS:
Drug: The TR group — Miscible liquid of triamcinolone acetonide and ropivacaine in this study will be peri-incisional scalp infiltration with 10ml ropivacaine 1% wt/vol, 0.25ml triamcinolone acetonide (40mg/ml), plus 10 ml saline miscible liquids for participants who will undergo elective craniotomy. Local infiltration of the study solution was performed by the neurosurgeon after induction of general anesthesia and intubation, once all equipment and catheters had been placed, during stable and steady state anesthetic conditions before skin incision. The solution was infiltrated with a 22-gauge needle introduced into the skin at a 45° angle throughout the entire thickness of the scalp along the planned incision site and the head-holder sites, by the same neurosurgeon. The total volume of the study solution used for each patient was determined by the neurosurgeon mainly based on the length of the incision and recorded by the investigator.
  Arms: The TR group
Drug: The R group — Miscible liquid of ropivacaine in this study will be peri-incisional scalp infiltration with 10ml ropivacaine 1% wt/vol, plus 10 ml saline miscible liquids for participants who will undergo elective craniotomy. Local infiltration of the study solution was performed by the neurosurgeon after induction of general anesthesia and intubation, once all equipment and catheters had been placed, during stable and steady state anesthetic conditions before skin incision. The solution was infiltrated with a 22-gauge needle introduced into the skin at a 45° angle throughout the entire thickness of the scalp along the planned incision site and the head-holder sites, by the same neurosurgeon. The total volume of the study solution used for each patient was determined by the neurosurgeon mainly based on the length of the incision and recorded by the investigator.
  Arms: The R group

SUMMARY:
Pain is common for the first 2 days after major craniotomy. A majority of patients would suffer from moderate-to-severe postoperative pain after undergoing craniotomy. Inadequate analgesia induced sympathetically mediated hypertension may lead to an increased risk for post-operative complications. Adequate pain control is essential for patients' prognosis and their postoperative life quality. Pain after craniotomy derives from the scalp and pericranial muscles. Local anesthetics administered around the incision have been performed clinically. However, some studies revealed that the analgesic effect of local anesthetics was not unsatisfactory due to its short pain relief duration. Pain is common for the first 2 days after major elective intracranial surgery, and the relatively short analgesic time of scalp infiltration does not seem to meet the requirements of craniotomy. Steroid such as triamcinolone acetonide as an adjuvant to local anesthetics intra-articular injected locally ameliorated pain intensity inarthroscopic knee surgery or total knee arthroplasty. However, there has not been reported about local application of triamcinolone acetonide on scalp infiltration. Thus, the investigators suppose that pre-emptive scalp infiltration with steroid (triamcinolone acetonide) plus local anesthetic (ropivacaine) could relieve postoperative pain after craniotomy in adults.

ELIGIBILITY:
Inclusion Criteria:

* Patients scheduled for elective craniotomy for resection of tumour under general anaesthesia;
* American Society of Anesthesiologists (ASA) physical status of I ,II or III;
* Participates with an anticipated fully recovery within 2 hours postoperatively;

Exclusion Criteria:

* History of craniotomy;
* Expected delayed extubation or no plan to extubate;
* Participants who cannot use a patient-controlled analgesia (PCA) device;
* Participants who cannot understand the instructions of a numeral rating scale (NRS) 35 before surgery;
* Extreme body mass index (BMI) (< 15 or > 35);
* Allergy to opioids, triamcinolone acetonide or ropivacaine;
* History of excessive alcohol or drug abuse, chronic opioid use (more than 2 weeks), or use of drugs with confirmed or suspected sedative or analgesic effects;
* History of psychiatric disorders, uncontrolled epilepsy or chronic headache;
* Pregnant or at breastfeeding;
* Symptomatic cardiopulmonary, renal, or liver dysfunction or history of diabetes;
* Preoperative Glasgow Coma Scale< 15;
* Suspicion of intracranial hypertension;
* Peri-incisional infection;
* Participants who have received radiation therapy and chemotherapy preoperatively or with a high probability to require a postoperative radiation therapy and chemotherapy according to the preoperative imaging.

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 110 (Actual)
Dates: Start 2023-10-07 (Actual); Primary Completion 2023-12-31 (Actual); Study Completion 2023-12-31 (Actual)

PRIMARY OUTCOMES:
Cumulative sufentanil consumption within 48 hours postoperatively | Within 48 hours after the operation
  All participates will receive an electronic intravenous patient-controlled analgesia (PCA) device. Participates will be advised to push the analgesic demand button if they feel pain.

SECONDARY OUTCOMES:
The first time to press the patient-controlled analgesia button | Within 48 hours after the operation
  The first time that the participants press the patient-controlled analgesia button.
The total times that participants press patient-controlled analgesia button | Within 48 hours postoperatively
  The total times that participants press patient-controlled analgesia button including effective presses and ineffective presses.
Numerical rating scale (NRS) | At 2 hours, 4 hours, 8 hours, 24 hours, 48 hours, 72 hours, 1 week, 2 weeks, 1 month,
  Pain will be assessed after surgery by numerical rating scale (0 indicates no pain, 10 indicates the most severe pain imaginable).
Postoperative nausea and vomiting | At 2 hours, 4 hours, 8 hours, 24 hours, 48 hours after surgery
  Postoperative nausea and vomiting (PONV) was rated by participates as: 0, absent; 1, nausea not requiring treatment; 2, nausea requiring treatment; and 3, vomiting.
The times of emergency reducing blood pressure after the operation | Within 48 hours after the operation
  The criteria for treatment is determined by the participant's surgeon in charge.The times of emergency reducing blood pressure will be recording by the investigator.
The total consumption of opioids during the operation | During procedure
  The total consumption of opioids during the operation
The length of stay | Approximately 2 weeks after the surgery
  The duration of hospitalization after the operation
Wound Healing Score | At 1 month after surgery
  Skin Healing 1: fully healed; 2: ≤3 cm in total not healed; 3: >3 cm not healed; 4: areas of necrosis ≤3 cm; 5: areas of necrosis >3 cm Infection 1: none; 2: ≤0.5-cm margin of redness; 3: more redness or superficial pus; 4: deep infection; not applicable Hair Regrowth 1: even regrowth along wound; 2: ≤3 cm not regrowing; 3: >3-6 cm not regrowing; 4: >6 cm not regrowing; not applicable

CONTACTS AND LOCATIONS:
Overall Officials: Fang Luo, M.D., Principal Investigator — Beijing Tiantan Hospital
Locations (1):
- Beijing Tiantan Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: Yes

REFERENCES:
- [Background] Gottschalk A, Berkow LC, Stevens RD, Mirski M, Thompson RE, White ED, Weingart JD, Long DM, Yaster M. Prospective evaluation of pain and analgesic use following major elective intracranial surgery. J Neurosurg. 2007 Feb;106(2):210-6. doi: 10.3171/jns.2007.106.2.210. PMID 17410701
- [Background] Dunn LK, Naik BI, Nemergut EC, Durieux ME. Post-Craniotomy Pain Management: Beyond Opioids. Curr Neurol Neurosci Rep. 2016 Oct;16(10):93. doi: 10.1007/s11910-016-0693-y. PMID 27604271
- [Background] Chaki T, Sugino S, Janicki PK, Ishioka Y, Hatakeyama Y, Hayase T, Kaneuchi-Yamashita M, Kohri N, Yamakage M. Efficacy and Safety of a Lidocaine and Ropivacaine Mixture for Scalp Nerve Block and Local Infiltration Anesthesia in Patients Undergoing Awake Craniotomy. J Neurosurg Anesthesiol. 2016 Jan;28(1):1-5. doi: 10.1097/ANA.0000000000000149. PMID 25493926
- [Background] Penning LI, de Bie RA, Walenkamp GH. Subacromial triamcinolone acetonide, hyaluronic acid and saline injections for shoulder pain an RCT investigating the effectiveness in the first days. BMC Musculoskelet Disord. 2014 Oct 23;15:352. doi: 10.1186/1471-2474-15-352. PMID 25341673
- [Background] Wang JJ, Ho ST, Lee SC, Tang JJ, Liaw WJ. Intraarticular triamcinolone acetonide for pain control after arthroscopic knee surgery. Anesth Analg. 1998 Nov;87(5):1113-6. doi: 10.1097/00000539-199811000-00024. PMID 9806691
- [Background] Sean VW, Chin PL, Chia SL, Yang KY, Lo NN, Yeo SJ. Single-dose periarticular steroid infiltration for pain management in total knee arthroplasty: a prospective, double-blind, randomised controlled trial. Singapore Med J. 2011 Jan;52(1):19-23. PMID 21298236
- [Background] Wesley CK, Teo LH, Xu T, Unger RH, Unger WP. The influence of peri-incisional triamcinolone acetonide injection on wound edge apposition. J Dermatolog Treat. 2014 Aug;25(4):345-9. doi: 10.3109/09546634.2012.755253. Epub 2013 Feb 3. PMID 23210735